CLINICAL TRIAL: NCT05342896
Title: Effect of Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Plus Forest Bathing (FB) on Blood Pressure and Cognitive Health for Those Who Are Aged 50 and Above With Hypertension
Brief Title: Effect of Mediterranean-DASH Intervention for Neurodegenerative Delay Plus Forest Bathing
Acronym: MINDdiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Queenie Law Pui Sze, Associate Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HE-NHS2021/02
Record Dates: First submitted 2021-12-06; First posted 2022-04-25 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: High Blood Pressure
Keywords: High Blood Pressure; MIND diet; Forest Bathing
MeSH Terms: conditions — Hypertension | interventions — Forest Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It will be a single-blind trial; only the assessors will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIND diet intervention (Experimental): 3-month intervention of dietary counseling to adhere to the MIND diet
  Interventions: Behavioral: MIND diet
- MIND-plus-FB intervention (Experimental): 3-month intervention of dietary counseling to adhere to the MIND diet plus Forest Bathing intervention
  Interventions: Behavioral: Mind diet plus Forest Bathing
- Control group (No Intervention): For the control group, the participants will be received routine care.

INTERVENTIONS:
Behavioral: MIND diet — MIND diet intervention will be a 3-month nutrition programme consisting of 4 face-to-face nutrition counselling sessions (one session per week, 60 min per session) in the activity room of each participating community centre. All intervention sessions will be conducted by a registered nutritionist and trained student helpers. In the nutrition sessions, the participants will learn to modify their diet to meet MIND diet guidelines.
  Arms: MIND diet intervention
Behavioral: Mind diet plus Forest Bathing — MIND diet intervention will be a 3-month nutrition programme consisting of 4 face-to-face nutrition counselling sessions (one session per week, 60 min per session) in the activity room of each participating community centre. All intervention sessions will be conducted by a registered nutritionist and trained student helpers. In the nutrition sessions, the participants will learn to modify their diet to meet MIND diet guidelines. Forest Bathing will be another session per week, 2 hours forest bathing sessions on 4-consecutive weekends in a country park at daytime with sunny, cloudy or drizzling conditions. The walking distance for each forest bathing is one to two kilometres. The coach-to-participant ratio is approximately 1:16. Participants will then be required to self-practice 2h FB in the country park at daytime at the weekends of 8th week and 12th week of the intervention.
  Arms: MIND-plus-FB intervention

SUMMARY:
This proposed study will be the first to investigate the effect of the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Plus Forest Bathing (FB) on blood pressure (BP) and cognitive health for those who are aged 50 and above with hypertension. Hypertension is a major public health issue, and four developments make this research study remarkably important.

It is well-documented the Mediterranean diet and Dietary Approach to Stop Hypertension (DASH) diet have demonstrated efficacy for improving cardiovascular and cognitive health. The Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet is a hybrid of the Mediterranean and DASH diets. FB promotes relaxation by inducing the activity of the parasympathetic nervous system, which decrease Heart rate and BP. The initial quantitative phase of the study, a three-arm RCT will be conducted to examine the effects of MIND, MIND plus FB and usual care as control on hypertension. The subsequent qualitative phase in-depth focus group interview is to explore the barriers and facilitators of MIND diet uptake and FB. The participants will include older HK Chinese adults who meet the criteria for hypertension stage 1 and stage 2 of the AHA. The primary outcomes are systolic BP and the secondary outcomes are point of care test of lipid panel, cognitive function, waist-to-hip ratio, body fat percentages and body mass index. The outcome measurements will be recorded before the interventions (T0), immediately after the 4-week face-to-face intervention (T1) and 12-week after 3-month intervention (T2). A total of 48 those who are aged 50 and above with hypertension will be recruited from community centres in Hong Kong to Randomized Controlled Trial and 10 participants differing in levels of compliance to MIND and FB will be purposively selected for face-to-face semi-structured focus group interviews.

DETAILED DESCRIPTION:
Research aim

1. This study will aim to investigate the effect of MIND and MIND plus FB on hypertension.
2. To examine the effect of MIND alone on hypertension by controlling other covariates.
3. To describe the perceived capability, opportunity, and motivation to the uptake of the MIND and FB.
4. To explore the barriers and facilitators to the MIND and FB.

The MIND-FB is proposed in response to (i) high BP is the one of important risk factors for chronic diseases. (ii) although there is robust evidence to show that the important of lowering BP to reduce chance of getting cardiovascular morbidity and mortality, the global burden of hypertension is still increasing. The objectives of MIND-FB are to perform high quality research focused on those who are aged 50 and above, novel transdisciplinary approaches to ensure the building capacity of public health workforce to deliver quality lifestyle modification intervention to control BP of those who are aged 50 and above.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 and above;
* Chinese ethnicity;
* ability to speak and understand Chinese;
* fulfilment of the AHA criteria for stage 1 and stage 2 hypertension; and
* who could walk independently

Exclusion Criteria:

* have allergy to more than one type of food (nuts, berries, olive oil, or fish);
* participation in any dietary or relaxation programme within the past 3 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Blood pressure | Three months
  By systolic blood pressure, measured by a digital automatic device

SECONDARY OUTCOMES:
Change in lipid panel of HDL cholesterol, triglycerides and LDL cholesterol | Three months
  By point of care test (POCT) of lipid panel (HDL-cholesterol, triglycerides and LDL-cholesterol)
Change in body fat percentages | Three months
  By body fat percentages, measured by bioelectrical impedance analysis
Change in cognitive function | Three months
  By cognitive function, measured by Hong Kong version of the Montreal Cognitive Assessment, cut-off score of 21/22 after adjustment of education level is recommended as indication for further evaluation of cognitive impairment and dementia. Lower scores mean worse outcome. The minimum score is 0 and maximum score is 30.
Change in waist circumference | Three months
  By waist circumference, measured by tape meter between the lower rib and iliac crest
Change in diet scores | Three months
  By diet scores, measured by total scores using predefined criteria of MIND diet. A value of 0.0, 0.5, or 1.0 is assigned to each food group. For high intake of brain healthy food group, participants will receive a score of 1 and the score is reversed for unhealthy food group. The total MIND diet score will be computed by summing all food groups eaten, with a maximum score of 15 representing the highest adherence to the MIND diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Queenie Law, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Will be shared by completion of data
Supporting Information: Study Protocol
Time Frame: June 2022
Access Criteria: Pilot result will be published in journal article

REFERENCES:
- [Background] 1. Morris M C., Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett, DA, & Aggarwal N T. MIND diet slows cognitive decline with aging. Alzheimer's and Dementia. 2015. 11(9): 1015-1022. 2. Morris MC, Tangney CC, Wang Y, Sacks FM, Bennett DA, & Aggarwal NT. MIND diet associated with reduced incidence of Alzheimer's disease. Alzheimer's and Dementia. 2015. 11(9): 1007-1014. 3. Aminianfar A, Hassanzadeh Keshteli A, Esmaillzadeh A, & Adibi P. Association between adherence to MIND diet and general and abdominal obesity: A cross-sectional study. Nutrition Journal. 2020. 19(1): 1-9. 4. Arjmand G, Abbas-Zadeh M, & Eftekhari MH. Effect of MIND diet intervention on cognitive performance and brain structure in healthy obese women: A randomized controlled trial. In bioRxiv. bioRxiv. 2020.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT05342896/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT05342896/ICF_001.pdf